CLINICAL TRIAL: NCT02212860
Title: Clinical Trial to Evaluate Single Dose Versus Three Doses of Stereotactic Radiation Therapy (SBRT) Prior to Surgery for Early Stage Breast Carcinoma: SIGNAL 2.0 (Stereotactic Image-Guided Neoadjuvant Ablative Radiation Then Lumpectomy) Trial
Brief Title: Stereotactic Image-Guided Neoadjuvant Ablative Radiation Then Lumpectomy
Acronym: SIGNAL 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Weill Medical College of Cornell University (Other); Sunnybrook Health Sciences Centre (Other); Ontario Institute for Cancer Research (Other)
Responsible Party: Principal Investigator, Muriel Brackstone, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SIGNAL
Record Dates: First submitted 2014-08-05; First posted 2014-08-08 (Estimated); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Early Stage Breast Carcinoma
Keywords: neoadjuvant; radiation; breast; cancer; hypofractionation; stereotactic; preoperative
MeSH Terms: conditions — Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Single Fraction (Experimental): Stereotactic neoadjuvant ablative radiation give in one single dose of 21 Gy. Lumpectomy to follow within 14-20 from radiation treatment date.
  Interventions: Radiation: Stereotactic Body Radiation Then Surgery
- Three Fractions (Experimental): Stereotactic neoadjuvant ablative radiation give in three doses of 10 Gy (30 Gy given in 3 fractions, one treatment every second business day). Lumpectomy to follow within 14-20 days from last radiation treatment.
  Interventions: Radiation: Stereotactic Body Radiation Then Surgery

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Then Surgery — Stereotactic image-guided neoadjuvant ablative radiation (randomized to single dose of 21 Gy or three 10 Gy doses) followed by lumpectomy for early stage breast carcinoma
  Other Names: Neoadjuvant radiation

SUMMARY:
Radiation therapy after surgery to remove breast cancer improves control of the breast cancer. Standard therapy after breast conservation surgery is five to six weeks of radiation to the entire breast.

This clinical trial will evaluate the effectiveness of conformal radiation therapy delivered only to the area in the breast where the lumpectomy will be performed.

This study will determine if radiation therapy delivered in this manner will prevent the cancer from coming back and eliminate the need for five to six weeks of radiation. Eligible participants will be randomized to one of two arms; Arm 1 which is comprised of one neoadjuvant radiation treatment, or Arm 2 which is comprised of three neoadjuvant radiation treatments.

The study will also gather information about the safety and effects (good and bad) this radiation has, the immune priming effects of this radiation, and on patient satisfaction with the appearance of the breast.

DETAILED DESCRIPTION:
Our proposal represents the convergence of several recent developments in the treatment of patients with low-risk carcinoma of the breast. For the selected subset of patients with low-risk disease, it appears that intra-operative radiotherapy with a single fraction leads to acceptable clinical outcomes in terms of local control, overall survival and toxicity. There have also been a few Phase I dose escalation trials demonstrating safety with single fraction breast radiation.

In this study, we propose the delivery of radiotherapy using stereotactic body radiation therapy in two different regimens; a single 21 Gy fraction, or 3 10Gy fractions. Radiation will be delivered using Volumetric-modulated arc therapy (VMAT), planned on coregistered MRI (with a subset having a 3T PET-MRI) and CT imaging, and delivered prone. Our approach will potentially have numerous benefits, including significantly shortened treatment time, convenience and potentially reduced health care costs. It would significantly improve the quality of life of many patients.

This study will also provide a unique opportunity for pathologic assessment of the impact of radiation at a microscopic level and on tumour and immune markers without the confounding impact of systemic treatments, comparing pre- to post-radiation biopsy specimens for imaging and histologic predictors of radiation sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 50 years and postmenopausal
* Tumor size < 3cm on pre-treatment imaging
* Any grade of disease, estrogen receptor (ER) positive
* Unicentric/unifocal disease
* Invasive ductal carcinoma or other favorable subtypes of epithelial breast malignancy (lobular, medullary, papillary, colloid, mucinous, or tubular) .
* Clinically node-negative (based upon pre-treatment physical examination and/or axillary ultrasound).
* Surgical expectation that a > 2mm margin can be obtained.
* Lesion is 1 cm or greater from the skin surface.
* Able to have surgery within 14-20 days of radiation therapy.
* Able to lie comfortably in the prone position with arms raised above the head for extended periods of time.

Exclusion Criteria:

* Previous RT to the same breast
* Evidence of suspicious diffuse microcalcifications in the breast prior to the start of radiation.
* Local metastatic spread into ipsilateral axilla and/or supraclavicular region and/or neck nodes and/or internal mammary nodes diagnosed on clinical examination or any imaging assessment (unless such sites can be confirmed as negative following biopsy)
* Distant metastases
* Involvement of contralateral axillary, supraclavicular, infraclavicular or internal mammary nodes (unless there is histologic confirmation that these nodes are negative)
* Prior non-hormonal therapy or radiation therapy for the current breast cancer
* Patients with Paget's disease of the nipple.
* Skin involvement, regardless of tumor size.
* Patients with a breast technically unsatisfactory for radiation therapy.
* Inability to lie prone with arms raised above head for extended periods of time.
* Patients not appropriate for breast conserving surgery due to expectation of poor cosmetic result, even without RT
* Collagen vascular disease (particularly lupus, scleroderma, dermatomyositis)
* Inability or unwillingness to provide informed consent.
* Any other malignancy at any site (except non-melanomatous skin cancer) < 5 years prior to study enrollment
* Patients who are pregnant or lactating

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-04-27 (Actual); Primary Completion 2021-04-23 (Actual); Study Completion 2024-04 (Actual)

PRIMARY OUTCOMES:
Immune priming will be measured | 1.5 years
  Immune priming effects of both treatment arms will be evaluated by quantifying tumour infiltrating lymphocytes (CD8) into tumour specimen, as well as the expression of immune markers (PDL1, Fox3) and immune panel in blood (CD4, CD8, neutrophil, and macrophage counts).
Angiogenesis will be measured | 1.5 years
  Angiogenesis will be examined using the CD31 or VEGF-a cell markers
Proliferation markers will be measured | 1.5 years
  Proliferation will be examined using the Ki67 marker, hypoxia will be examined using the Carbonic Anhydrase 9 (CAH IX), or HIF1/HIF2 markers, apoptosis will be examined using the Caspase-3, or Tunnel markers, invasion will be analyzed using the vimentin, or SDF1-a markers.
Hypoxia markers will be measured | 1.5 years
  Hypoxia will be examined using the Carbonic Anhydrase 9 (CAH IX), or HIF1/HIF2 markers, apoptosis will be examined using the Caspase-3, or Tunnel markers, invasion will be analyzed using the vimentin, or SDF1-a markers.
Apoptosis markers will be measured | 1.5 years
  Apoptosis will be examined using the Caspase-3, or Tunnel markers, invasion will be analyzed using the vimentin, or SDF1-a markers.
Invasion markers will be measured | 1.5 years
  Invasion will be analyzed using the vimentin, or SDF1-a markers.
Toxicity resulting from radiation treatment | 1.5 years
  Toxicity resulting from radiation treatment will be collected and graded according to the Common Terminology Criteria for Adverse Events, version 4.0

SECONDARY OUTCOMES:
Cosmesis of the treated breast | 1.5 years
  cosmetic result of treated breast as judged by the patient, surgeon, and radiation oncologist. Patients will self-assess cosmesis using the Modified Harvard-Harris Cosmetic Scale. The surgeon and radiation oncologist will assess cosmesis using photographs and the Modified Harvard-Harris Cosmetic Scale.
Disease-Free Survival | 8.5 years
  Disease recurrences will be recorded. Any tumor recurrence or death is considered a treatment failure.
Mastectomy-Free Survival | 8.5 years
  All surgical interventions will be recorded. Mastectomy and death will be considered treatment failures.
Overall Survival | 8.5 years
  Death from any cause is considered a treatment failure.

CONTACTS AND LOCATIONS:
Overall Officials: Muriel Brackstone, MD, PhD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- London Regional Cancer Program of the Lawson Health Research Institute, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No